CLINICAL TRIAL: NCT06321796
Title: Microbiota Transfer Therapy for Children and Adults With Both Pitt Hopkins Syndrome and Gastrointestinal Disorders: MTP-101 P
Brief Title: Microbiota Transfer Therapy for Children and Adults With Both Pitt Hopkins Syndrome and Gastrointestinal Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gut-Brain-Axis Therapeutics Inc. (Other)
Collaborators: Pitt Hopkins Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WCG IRB Protocol #20235847
Record Dates: First submitted 2024-03-07; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pitt Hopkins Syndrome
Keywords: Microbiota Transfer Therapy; Fecal Transplant; Fecal Microbiota Transplant; Intestinal Microbiota
MeSH Terms: conditions — Pitt-Hopkins syndrome | interventions — Vancomycin; magnesium citrate; Antacids

STUDY DESIGN:
Intervention Model Description: Part 1: Randomized, Double-Blinded, Placebo-Controlled Treatment (14 weeks) Part 2: Open-Label Observation and Cross-over or Treatment Part 3: Follow Up (Group B Only)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Treatment (Experimental): Part 1: Blinded Treatment (14 weeks)
  Vancomycin, Magnesium Citrate, Antacid, MTP-101P
  Interventions: Combination Product: MTP-101P; Combination Product: Vancomycin; Combination Product: Magnesium Citrate; Combination Product: Antacid
- Group B: Placebo (Placebo Comparator): Part 1: Blinded Placebo (14 weeks)
  Placebo Vancomycin, Real Magnesium Citrate, Real Antacid, Placebo MTP-101P
  Interventions: Combination Product: Magnesium Citrate; Combination Product: Antacid; Combination Product: Placebo MTP-101P; Combination Product: Placebo Vancomycin

INTERVENTIONS:
Combination Product: MTP-101P — MTP-101P is comprised of standardized dose of total fecal microbiota purified from the stool of healthy donors. Donors are carefully screened via health status questionnaires, physical examinations, reviews of comprehensive medical history, clinical laboratory evaluations, serologic and genomic tests for infectious diseases and metabolic health, and stool-related pathogen testing. The material from the donors is purified to remove the majority of non-bacterial material, washed, lyophilized, and provided to the patient in a sachet contained within a mixing bottle.
  Duration: 12.5 Weeks
  Arms: Group A: Treatment
Combination Product: Vancomycin — Oral vancomycin is an antibiotic used for treating C. difficile-associated diarrhea and staphylococcal-induced enterocolitis.
  Duration: 10 Days
  Arms: Group A: Treatment
Combination Product: Magnesium Citrate — Magnesium citrate is a common over-the-counter laxative and bowel cleanse.
  Duration: 1 Day
Combination Product: Antacid — The antacid will be aluminum/magnesium hydroxide, 1x/day, 5 minutes before the MTP-101P. Each 5 ml consists of Aluminum Hydroxide - 200 mg, Magnesium Hydroxide - 200 mg, and Simethicone - 20 mg. If some participants cannot tolerate the aluminum/magnesium hydroxide, we will allow calcium carbonate alternatives equivalent in acid neutralizing capacity.
  Duration: 12.5 weeks
Combination Product: Placebo MTP-101P — The same packaging will be used as for MTP-101P, but the sachets will contain a freeze-dried mixture of normal saline containing 10% Trehalose.
  Duration: 12.5 weeks
  Arms: Group B: Placebo
Combination Product: Placebo Vancomycin — Same packaging and liquid carrier and flavoring used as for the oral vancomycin, but no vancomycin.
  Duration: 10 days
  Arms: Group B: Placebo

SUMMARY:
The investigators propose to investigate Microbiota Transfer Therapy (MTT) for treating patients with Pitt-Hopkins Syndrome (PTHS) and gastrointestinal problems (constipation, bloating, abdominal pain). MTT involves a combination of 10 days of oral vancomycin (an antibiotic to kill pathogenic bacteria), followed by 1 day of bowel cleanse using magnesium citrate, followed by 4 days of high dose MTP-101P with an antacid, followed by 12 weeks of a lower maintenance dose of MTP-101P with an antacid.

DETAILED DESCRIPTION:
For children 5-17 years old and adults 18-55 years old with Pitt-Hopkins Syndrome (PTHS) and Gastrointestinal (GI) problems who have attempted two standard-of-care (SOC) GI treatments with no alleviation of symptoms. This is a Phase 2 clinical trial that will evaluate the safety, tolerability, and efficacy of a powder version of Microbiota Transfer Therapy (MTT) called MTP-101P. The three parts of this trial are described below.

Part 1: Placebo-Controlled Treatment (14 Weeks) The trial will begin with a randomized, double-blind, placebo-controlled trial which will include a 10-day treatment with oral vancomycin (or placebo), then 1 day of magnesium citrate to cleanse the bowel of vancomycin and bacteria/feces (all participants, since its bowel-emptying effect cannot be blinded), followed by 4 days of initial high dose of MTP-101P taken daily 5 minutes after antacid, and then 12 weeks of a lower maintenance dose of MTP-101P taken daily 5 minutes after an antacid.

Group A: Real Treatment vs. Group B: Placebo vancomycin, real magnesium citrate, placebo MTP-101P, real antacid.

Part 2: Open-Label Observation and Cross-Over (14 weeks) Group A: Observation over the next 14 weeks (no additional treatment). Group A completes the study at the end of part 2.

Group B: They will receive the same treatment that Group A received in part 1. This includes 10 days of vancomycin, magnesium citrate, and an initial high dose of MTP-101P for 4 days taken daily 5 minutes after an antacid, and then a lower dose of MTP-101P for 12 weeks taken daily 5 minutes after antacid.

Part 3: Follow Up Group B: There will be a follow-up evaluation 14 weeks post-treatment after the end of Part 2, to assess long-term efficacy and possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 5 to <18 years and adults ages 18 to < 55 years with Pitt Hopkins Syndrome (verified by genetic testing)
2. GI disorder as defined below that has lasted for at least 2 years.
3. No changes in medications, supplements, diet, or therapies in the 2 months prior to start of treatment, and no intention to change treatments during Part 1 (all participants) and Part 2 (group B) of the clinical trial. The only exception is GI medications, which may be reduced if symptoms reduce, and any changes during the study will be documented.
4. Review of last year of medical records by the study physician.
5. At least two previous trials of "standard of care" GI treatments that did not alleviate GI symptoms (constipation, diarrhea, bloating, gas, reflux, and/or abdominal pain). Standard of care treatments include laxatives, stool softeners, enemas, suppositories, or similar medications.

Exclusion Criteria:

1. Antibiotics in 2 months prior to start of treatment (topical antibiotics are allowed)
2. Probiotics in 2 months prior to start of treatment, or fecal transplant in last 12 months. Foods naturally containing probiotics such as yogurt are allowed.
3. Tube feeding may be an exclusion criterion if the participant requires an unusual diet such as a liquid diet with low fiber.
4. Current severe gastrointestinal problems that require immediate hospital treatment (life-threatening)
5. Ulcerative Colitis, Crohn's Disease, diagnosed Celiac Disease, Eosinophilic Gastroenteritis, or similar conditions
6. Unstable, poor health (based on study physician's opinion), or active malignancy or infection.
7. Recent or scheduled abdominal surgeries
8. Current participation in other clinical trials
9. Females who are pregnant or who are at risk of pregnancy and sexually active with a male partner without effective birth control. We will conduct a pregnancy test on all female participants 12 years and older as part of the screening and at each clinical visit.

   Males who are sexually active with a female partner without highly effective birth control (IUD or birth control hormones).
10. Allergy or intolerance to the study medications: vancomycin, magnesium citrate, milk powder with chocolate flavoring (which are included in MTP-101P), or the antacid.
11. Clinically significant abnormalities at baseline on the blood safety tests, and confirmed on a second test. The tests include Comprehensive Metabolic Panel, and Complete Blood Count with Differential. Note that some abnormalities may occur due to PTHS, so only those likely to significantly increase risk in this study would be grounds for exclusion, at the discretion of the study physician. See detailed discussion at the end of this section on Interpreting Laboratory Results. re. Eligibility for Admission to Study.
12. Evidence of significant impairment of immune system, or taking medications that can compromise the immune system, and thus increase risk if exposed to multiple-drug resistant bacteria.
13. Substantially decreased kidney function, as evidenced by estimated glomerular filtration rate of <60 mL/min/1.73 m2. This is not normally reported for children on standard laboratory metabolic panels, so in those cases we will use the National Kidney Foundations Pediatric Glomerular filtration rate (GFR) Calculator to calculate the pediatric GFR based on age/height, the Blood urea nitrogen (BUN) and serum creatinine from our standard Comprehensive Metabolic Panel (CMP). [https://www.kidney.org/professionals/kdoqi/gfr_calculatorped] This calculator uses the Creatinine-based "Bedside Schwartz" equation (2009) that seems to be the most commonly used calculation for this purpose.
14. Participants who are breastfeeding.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Daily Stool Record (DSR) | Baseline (for 14 days pre-treatment) vs End of Treatment (Days 82-95 of treatment).
  Participants will report the number of abnormal events during a 14 day period. An event includes no bowel movement during 1 day, unusually hard stool (Bristol Stool Form type 1-2), unusually soft stool (Bristol Stool Form type 6-7), four or more bowel movements in 1 day, abdominal pain, or use of GI medication. The units are number of events regardless of type of event.
Safety Measures (Adverse Events) | Days 0 to 99 of treatment
  Safety will be assessed based on the number of adverse events during treatment for each group (Group A and Group B). Units are number of adverse events.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | Baseline (pre-treatment) vs End of Treatment (After 95 days of treatment)
  An assessment of GI symptoms based on 15 questions, which are then scored in five domains (abdominal pain, reflux, indigestion, diarrhea, and constipation). Symptoms are rated on a 7-point Likert scale including no discomfort at all (1), slight discomfort (2), mild discomfort (3), moderate discomfort (4), moderately severe discomfort (5), severe discomfort (6), and very severe discomfort (7).
Clinical Global Impression - Gastrointestinal (CGI-GI) | Baseline (pre-treatment) vs End of Treatment (After 99 days of treatment)
  This assessment is conducted by the study physician and assess the severity of GI symptoms on a 7-point scale. The severity scale rates the severity of the patient's illness including normal, not at all ill (1), borderline mentally ill (2), mildly ill (3), moderately ill (4), markedly ill (5), severely ill (6), among the most extremely ill patients (7).
Clinical Global Impression - Pitt Hopkins (CGI-PTHS) | Baseline (pre-treatment) vs End of Treatment (After 99 days of treatment).
  This assessment is conducted by the study physician and assess the severity of Pitt Hopkins Symptoms on a 7-point scale. The severity scale rates the severity of the patient's illness including normal, not at all ill (1), borderline mentally ill (2), mildly ill (3), moderately ill (4), markedly ill (5), severely ill (6), among the most extremely ill patients (7).
Parent Global Impressions - Pitt Hopkins: Change in Symptoms (PGI-PTHS-2-Change) | End of Treatment (After 95 days of treatment)
  An assessment of Pitt Hopkins Syndrome symptoms that rates the change in symptom severity since the start of treatment. Symptom severity is rated on a 7-point scale including much worse (-3), somewhat worse (-2), slightly worse (-1), no change (0), slightly better (1), somewhat better (2), and much better (3).
Gastrointestinal Symptoms common in Pitt Hopkins (GI-PTHS) | Baseline (pre-treatment) vs End of Treatment (After 95 days of treatment)
  Assess common symptoms in Pitt Hopkins, including 2 questions about toilet training, a question about GI feeding tubes, and 7 questions about current GI symptom severity including constipation, diarrhea, gas, bloating, pain, reflux/heartburn/regurgitation and vomiting. Symptoms are rated on a 7-point scale from none to extremely severe.
Revised Face Legs Activity Crying Consolability Pain Questionnaire (FLACC) | Baseline (pre-treatment) vs End of Treatment (After 95 days of treatment)
  Modified from the original FLACC for children with cognitive impairment (Malviya et al., 2006). Assess pain in five areas (Face, Legs, Activity, Crying, Consolability) using a three-point scale for each area, resulting in a total FLACC pain scale ranging from zero to 10.
National Survey on treatment Effectiveness for Autism (NSTEA) - Overall Benefit | End of Treatment (After 95 days of treatment)
  Assess the effectiveness of MTT on overall benefit (no benefit (0)/slight benefit(1)/moderate benefit (2)/good benefit (3)/great benefit (4)).
National Survey on treatment Effectiveness for Autism (NSTEA) - Overall Adverse E | End of Treatment (After 95 days of treatment)
  Assess the effectiveness of MTT on overall adverse effects of treatment (no adverse effects (0)/mild adverse effects (1)/moderate adverse effects (2)/severe adverse effects (3)).

CONTACTS AND LOCATIONS:
Locations (1):
- Autism/Asperger's Research Group at Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No